CLINICAL TRIAL: NCT00174070
Title: Etiologies and Outcomes Analysis of Acute Respiratory Failure in Community
Brief Title: Etiologies and Outcomes of Acute Respiratory Failure in Community
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700726
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-11-03 (Estimated); Status verified 2005-07

CONDITIONS: Respiratory Failure
Keywords: Respiratory failure; Community
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Acute respiratory failure (ARF) remains a common reason for admission to the intensive care unit (ICU). ARF to be present in 32% of patients on ICU admission, with a further 24% of patients developing ARF during the ICU stay. A total of 56% of all ICU admissions for a length of >48 h had ARF at some point during their stay. The incidence of ARF was from 88.6 to 137.1 hospitalizations per 100,000 residents. The incidence of ARF was found to increase nearly exponentially with each decade until age 85 years. However, there is still paucity data about etiology and outcomes of acute respiratory failure happened in community.

Mortality of ARF in critically ill patients is between 40% and 65%. Independent hazards for ARF mortality include older age, severe chronic co-morbidities (HIV, active malignancy, cirrhosis), certain precipitating events (trauma, drug overdose, bone marrow transplant), and multiple organ system failure (MOSF) [7-9]. Mortality has also been associated with acute lung injury or bilateral infiltrates on chest radiograph, and with an elevated acute physiology score.

ARF patients form a large percentage of all ICU admissions and many factors might influence the final outcomes. With the high incidence of ARF in ICU, any improvement in the outcome of such population is likely to have marked effect on intensive care resource allocation. We wish this study may provide some valuable information about acute respiratory failure in community and improve the outcome of these patients.

DETAILED DESCRIPTION:
Acute respiratory failure (ARF) remains a common reason for admission to the intensive care unit (ICU). ARF to be present in 32% of patients on ICU admission, with a further 24% of patients developing ARF during the ICU stay [1]. A total of 56% of all ICU admissions for a length of >48 h had ARF at some point during their stay [1]. The incidence of ARF was from 88.6 to 137.1 hospitalizations per 100,000 residents [2, 3]. The incidence of ARF was found to increase nearly exponentially with each decade until age 85 years. However, there is still paucity data about etiology and outcomes of acute respiratory failure happened in community.

Mortality of ARF in critically ill patients is between 40% and 65% [2, 4-6]. Independent hazards for ARF mortality include older age, severe chronic co-morbidities (HIV, active malignancy, cirrhosis), certain precipitating events (trauma, drug overdose, bone marrow transplant), and multiple organ system failure (MOSF) [7-9]. Mortality has also been associated with acute lung injury or bilateral infiltrates on chest radiograph [6], and with an elevated acute physiology score [9-10].

ARF patients form a large percentage of all ICU admissions and many factors might influence the final outcomes. With the high incidence of ARF in ICU, any improvement in the outcome of such population is likely to have marked effect on intensive care resource allocation. We wish this study may provide some valuable information about acute respiratory failure in community and improve the outcome of these patients.

References:

1. Vincent JL, Akca S, De Mendonca A, et al: The epidemiology of acute respiratory failure in critically ill patients. Chest 2002; 121:1602-1609
2. Lewandowski K, Mets J, Deutschmann H, et al. Incidence, severity, and mortality of acute respiratory failure in Berlin, Germany. Am J Respir Crit Care Med 1995; 151:1121-1125
3. Behrendt CE. Acute respiratory failure in the United States: incidence and 31-day survival. Chest 2000; 118:1100-1105
4. Miberg JA, Davis DR, Steinberg KP, et al. Improved survival of patients with acute respiratory distress syndrome (ARDS): 1983-1993. JAMA 1995; 273:306-309
5. Doyle LA, Szaflarski N, Modin GW, et al. Identification of patients with acute lung injury: predictors of mortality. Am J Respir Crit Care Med 1995; 152:1818-1824
6. Luhr OR, Antonsen K, Karlsson M, et al. Incidence and mortality after acute respiratory failure and acute respiratory distress syndrome in Sweden, Denmark, and Iceland: The ARF Study Group. Am J Respir Crit Care Med 1999; 159:1849-1861
7. Vasilyev S, Schaap RN, Mortensen JD. Hospital survival rates of patients with acute respiratory failure in modern respiratory intensive care units. Chest 1995; 107:1083-1088
8. Stauffer JL, Fayter NA, Graves B, et al. Survival following mechanical ventilation for acute respiratory failure in adult men. Chest 1993; 104:1222-1229
9. Knaus WA. Prognosis with mechanical ventilation: the influence of disease, severity of disease, age, and chronic health status on survival from an acute illness. Am Rev Respir Dis 1989; 140:S8-S13
10. Epstein SK, Vuong V. Lack of influence of gender on outcomes of mechanically ventilated medical ICU patients. Chest 1999; 116:732-739

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory failure with mechanical ventilation
* Respiratory failure happened within 48 hours after admission
* Age > 18 y/o

Exclusion Criteria:

* Pregnanacy
* Transfer from other hospital with mechanical ventilation
* Mechanical ventilation after scheduled operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-08; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Lin Hsu, MD, Principal Investigator — Physcian
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Vincent JL, Akca S, De Mendonca A, Haji-Michael P, Sprung C, Moreno R, Antonelli M, Suter PM; SOFA Working Group. Sequntial organ failure assessment. The epidemiology of acute respiratory failure in critically ill patients(*). Chest. 2002 May;121(5):1602-9. doi: 10.1378/chest.121.5.1602. PMID 12006450
- [Background] Lewandowski K, Metz J, Deutschmann C, Preiss H, Kuhlen R, Artigas A, Falke KJ. Incidence, severity, and mortality of acute respiratory failure in Berlin, Germany. Am J Respir Crit Care Med. 1995 Apr;151(4):1121-5. doi: 10.1164/ajrccm.151.4.7697241.
- [Background] Behrendt CE. Acute respiratory failure in the United States: incidence and 31-day survival. Chest. 2000 Oct;118(4):1100-5. doi: 10.1378/chest.118.4.1100. PMID 11035684
- [Background] Milberg JA, Davis DR, Steinberg KP, Hudson LD. Improved survival of patients with acute respiratory distress syndrome (ARDS): 1983-1993. JAMA. 1995 Jan 25;273(4):306-9. PMID 7815658
- [Background] Doyle RL, Szaflarski N, Modin GW, Wiener-Kronish JP, Matthay MA. Identification of patients with acute lung injury. Predictors of mortality. Am J Respir Crit Care Med. 1995 Dec;152(6 Pt 1):1818-24. doi: 10.1164/ajrccm.152.6.8520742.
- [Background] Luhr OR, Antonsen K, Karlsson M, Aardal S, Thorsteinsson A, Frostell CG, Bonde J. Incidence and mortality after acute respiratory failure and acute respiratory distress syndrome in Sweden, Denmark, and Iceland. The ARF Study Group. Am J Respir Crit Care Med. 1999 Jun;159(6):1849-61. doi: 10.1164/ajrccm.159.6.9808136. PMID 10351930
- [Background] Vasilyev S, Schaap RN, Mortensen JD. Hospital survival rates of patients with acute respiratory failure in modern respiratory intensive care units. An international, multicenter, prospective survey. Chest. 1995 Apr;107(4):1083-8. doi: 10.1378/chest.107.4.1083. PMID 7705120
- [Background] Stauffer JL, Fayter NA, Graves B, Cromb M, Lynch JC, Goebel P. Survival following mechanical ventilation for acute respiratory failure in adult men. Chest. 1993 Oct;104(4):1222-9. doi: 10.1378/chest.104.4.1222. PMID 8404197
- [Background] Knaus WA. Prognosis with mechanical ventilation: the influence of disease, severity of disease, age, and chronic health status on survival from an acute illness. Am Rev Respir Dis. 1989 Aug;140(2 Pt 2):S8-13. doi: 10.1164/ajrccm/140.2_Pt_2.S8. PMID 2669589
- [Background] Epstein SK, Vuong V. Lack of influence of gender on outcomes of mechanically ventilated medical ICU patients. Chest. 1999 Sep;116(3):732-9. doi: 10.1378/chest.116.3.732. PMID 10492280